CLINICAL TRIAL: NCT04981873
Title: Translation And Validation Of The Pelvic Floor Distress Inventory Short Form (PFDI-20) To Urdu Language
Brief Title: UrduTranslation And Validation Of The Pelvic Floor Distress Inventory Short Form (PFDI-20)
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/0839 Bakhtawar Aslam
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Pelvic Floor Disorders
Keywords: pelvic floor distress inventory; pelvic floor disorders; postmenupausal women
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To translate and culturally adapt PELVIC FLOOR DISTRESS INVENTORY SHORT FORM (PFDI-20) into Urdu and To evaluate the reliability and validity of Urdu version of Pelvic floor distress inventory (short form).Urdu is the national language of Pakistan. The PFDI-20 has not been translated into Urdu so far. In order to use in Urdu speaking people, it is necessary to translate and culturally adapt PFDI-20 into Urdu language, so that it can be better understood by this population.

DETAILED DESCRIPTION:
Pelvic floor disorders, which include urinary incontinence, fecal incontinence, and pelvic organ prolapse, are highly prevalent conditions in women, affecting overall, almost 25% of women in the United States Because there are different types of pelvic floor disorders (PFDs), symptoms of different PFDs can vary or overlap. For example, women with PFDs may feel: heaviness, fullness, pulling, or aching in the vagina that gets worse by the end of the day or is related to a bowel movement; See or feel a "bulge" or "something coming out" of the vagina, have difficulty starting to urinate or emptying the bladder completely, leak urine when coughing, laughing, or exercising, feel an urgent or frequent need to urinate, feel pain while urinating, leak stool or have difficulty controlling gas, have constipation and have difficulty making it to the bathroom in time PFDI-20 has been translated into many languages across the globe to check the validity, reliability and responsiveness of the scale, in their native languages.

A study was conducted to assess validity of PFDI-20 in Finnish by using Multistep translation method with sample size of 63, they found it a valid tool.

In Turkish language validity and reliability of this tool was addressed on larger number of women and was recommended as valid and reliable tool

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women aged 45 years and older, those who can read and understand Urdu language

Exclusion Criteria:

* Previous pelvic surgery, Malignant tumor, Cognitive impairment and Dementia

Min Age: 45 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — pelvic floor disorders are most common in females
Study Population: Menopausal women aged 45 years and over
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Translatin and validation of Pelvic floor distress inventory short form(PFDI-20) | 6 months
  The Pelvic Floor Distress Inventory-20 is to measure health related quality of life of females suffering from pelvic floor disorders. it contains 3 scales and total 20 questions.3 scales are Urinary distress inventory,Pelvic organ prolapse distress inventory and Colorectal-anal distress inventory.Each question indicate presence of symptom by marking YES/NO and further describes the degree of discomfort by 4 variables,NOT AT ALL,SOMEWHAT,MODERATELY and QUITE A BIT.

SECONDARY OUTCOMES:
reliability | 6 months
  To determine reliability of Pelvic floor distress inventory short form(PFDI-20) in (URDU) language. reliability refers to ability of a measure to produce same results administered at two or more intervals. Thus this will be test through test retest reliability

OTHER OUTCOMES:
validity | 6 months
  to determine the validity of translation of PFDI-20 in (URDU) language. Validity is defined as how accurate the results are. Thus this will be measured through various parameters

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, Principal Investigator — Riphah International University
Locations (1):
- Margalla general hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443
- [Background] Mattsson NK, Nieminen K, Heikkinen AM, Jalkanen J, Koivurova S, Eloranta ML, Suvitie P, Tolppanen AM. Validation of the short forms of the Pelvic Floor Distress Inventory (PFDI-20), Pelvic Floor Impact Questionnaire (PFIQ-7), and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) in Finnish. Health Qual Life Outcomes. 2017 May 2;15(1):88. doi: 10.1186/s12955-017-0648-2. PMID 28464936
- [Background] Kaplan PB, Sut N, Sut HK. Validation, cultural adaptation and responsiveness of two pelvic-floor-specific quality-of-life questionnaires, PFDI-20 and PFIQ-7, in a Turkish population. Eur J Obstet Gynecol Reprod Biol. 2012 Jun;162(2):229-33. doi: 10.1016/j.ejogrb.2012.03.004. Epub 2012 Apr 4. PMID 22480412